CLINICAL TRIAL: NCT04398784
Title: Effect of Whole Blueberry Powder Consumption on Depression: A Randomized, Double-blind, Placebo Controlled, Crossover Study
Brief Title: Effect of Whole Blueberry Powder Consumption on Depression in a Central Louisiana Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University, Baton Rouge (Other)
Collaborators: U.S. Highbush Blueberry Council (Other); Louisiana Health Care Practitioners, LLC (Unknown); Collective Healthcare Solutions, LLC (Unknown); uBiome, Inc. (Unknown)
Responsible Party: Principal Investigator, Joseph Francis, Ph.D, Professor, Louisiana State University, Baton Rouge
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 46680
Record Dates: First submitted 2020-03-29; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Depression; Depression, Anxiety; Inflammation
Keywords: depression; inflammation; anxiety; blueberries
MeSH Terms: conditions — Depression; Anxiety Disorders; Inflammation

STUDY DESIGN:
Intervention Model Description: This study will utilize a randomized, double-blind, placebo-controlled, crossover design. 60 participants with depression will be randomized into either the placebo first or blueberry first group. Randomization will be based on outcomes from behavioral measures (Major Depression Inventory and GAD-7) and a physiological measure (C-reactive protein levels) in appointment 0. The first arm will consist of 12 weeks of daily treatment and baseline (pre-intervention), mid-intervention and post-intervention assessments. Next there will be a four week washout period, after which patients will switch treatments, and the second arm will commence--identical to the first in structure. Further, the study is a repeated measures design with each participant's baseline measures serving as her or his own control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blueberry treatment and placebo powders have been supplied by the U.S. Highbush Blueberry Council; packets are labeled either alpha or omega. The treatment powder is a freeze-dried whole blueberry powder, and the placebo is a color- and flavor-matched powder which has been used in previous trials. Only an unblinded research assistant will have knowledge of which label corresponds to blueberry or placebo. That research assistant will be in charge of: (1) Before each appointment, distributing appropriate treatment or placebo packets into closable boxes with a number corresponding to each participant. Care-providers will give closed boxes to participants at the time of assessment. (2) Re-labeling all collected data and samples with a participant code number, and sorting into appropriate groups for analysis by blinded researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1-Blueberry First/Placebo First (Other): Participants will be randomly assigned into either blueberry-first treatment or placebo-first group.
  Interventions: Dietary Supplement: Freeze Dried Blueberry Powder - 71717; Dietary Supplement: USHBC Blueberry Placebo Formula #114
- 2-Crossover (Other): Participants who received blueberry treatment will switch to placebo and vice versa.
  Interventions: Dietary Supplement: Freeze Dried Blueberry Powder - 71717; Dietary Supplement: USHBC Blueberry Placebo Formula #114

INTERVENTIONS:
Dietary Supplement: Freeze Dried Blueberry Powder - 71717 — Single serve packets containing 22.5 grams of powdered freeze-dried whole blueberries; A mix of 2 species, Vaccinium virgatum (ashei)/Vaccinium corymbosum, provided by U.S Highbush Blueberry Council (USHBC). Powders are sealed in single serve packets to protect from light and moisture. Packets are refrigerated except for when distributed to participants; participants are asked to store packets in refrigerator until consumption.
  Other Names: Tifblue/Rubel 50/50 Blend
Dietary Supplement: USHBC Blueberry Placebo Formula #114 — Blueberry flavor- and color-matched placebo powder.

SUMMARY:
This pilot study aims to measure the effects of an intervention of 22.5 grams of freeze-dried whole blueberry powder in water drunk daily. Measures are on outcomes of depression, biological markers of inflammation and oxidative stress, and microbial populations in the intestines.

DETAILED DESCRIPTION:
A 29 week double-blind, placebo-controlled, crossover intervention assessing the effect of a blueberries on behavioral symptoms related to depression, biological markers of inflammation and oxidative stress, and gut microbiome measures. A total of 45 participants will be randomly assigned to either a blueberry-first or placebo-first group; participants will take 22.5 grams of either freeze-dried blueberry powder or matched placebo powder mixed with water daily for 12 weeks. This period is followed by a 4 week washout period at the beginning of which all participants will stop the assigned intervention. After this washout the participants will start their crossover intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a stable diagnosis of Major Depressive Disorder (>1 year prior to enrollment)
* Males and females 18-70 years of age
* Subjects with sleep disruptions
* Subjects currently prescribed to a non-antipsychotic mono-pharmacotherapies
* English speaking subjects only (all evaluations are in English)

Subjects with the following inflammatory disorders that exhibit low to moderate symptoms:

* Hypertension (mild=140/80-160/90; moderate= 160/90-180/100)
* Asthma (requiring 2 or fewer inhalations of rescue inhaler per day)
* Gastroesophageal reflux disease
* Irritable bowel syndrome (controlled, <3 bowel movements a day)
* Arthritis (controlled)
* Chronic stomach ulcers (controlled)
* Obesity BMI <40
* Chronic pain
* Fibromyalgia
* Chronic Fatigue Syndrome
* Type I or Type II diabetes (controlled)
* Subjects that are compliant with current treatment regimens and clinic appointments
* Subjects taking intermittent or infrequent doses of acetaminophen or NSAIDs
* Subjects who currently smoke or have a history of smoking

Exclusion Criteria:

Subjects with current diagnosis or history of the following conditions; or subjects currently on medication for any of the following conditions:

* Severe Cardiovascular disease; Heart attack/pacemaker
* Cancer
* Autoimmunity Disorders
* Crohn's Disease or Ulcerative Colitis
* Alzheimer's Disease
* Parkinson's Disease
* Multiple Sclerosis
* Uncontrolled Diabetes: Type I or II
* Severe irritable bowel disease (>3 stools per day)
* Hypertension (severe >180/100)
* Hypotension (<100/60)
* Epilepsy
* Autism Spectrum Disorder
* Schizophrenia
* Psychosis/Psychotic Symptoms
* Uncontrolled Hypo/Hyperthyroidism
* Women who are pregnant, nursing, lactating, or planning to become pregnant within timeline of study
* Subjects who are blind or deaf
* Subjects who are allergic to blueberries or other similar foods or drinks (e.g. wine), or subjects who are allergic to red or blue food dye agents
* Subjects who do not like the taste of blueberries
* Subjects who do not want to disclose information related to their Major Depressive Disorder
* Subjects who do not want to be subjected to blood draws
* Subjects who consume >4 cups of blueberries per week or other foods/drinks with significant polyphenol content
* Subjects supplementing with elderberry syrup >4 times per week
* Subjects who have a planned surgery during the timeline of the study
* Subjects prescribed to antipsychotics
* Subjects using acetaminophen or NSAIDS (drugs targeting pro-inflammatory paths) chronically or exceeding recommended daily doses
* Subjects chronically on Decadron, Dexamethasone, or Prednisone; or other oral steroids
* Subjects on any augmenting agents (the following is not an inclusive list):

Abilify (aripiprazole), Risperdal (risperidone), Zyprexa (olanzapine), Seroquel (quetiapine), Clozaril(clozapine), Symbyax (olanzapine/fluoxetine), Geodon (ziprasidone)

* Subjects supplementing with devil's claw, fenugreek, guar gum, Panax ginseng, and Siberian ginseng
* Subjects who have a history of suicidal ideation or suicide attempt
* Subjects with a history or record of physical violence toward self or others
* Subjects who will jeopardize their job if they miss work for appointments
* Subjects with a history of addiction, except cigarettes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Major Depression Inventory (MDI) | Day 1 of treatment intervention, before treatment consumption
  A brief (10-Item) behavioral survey for assessing clinical depression symptoms and severity; can confirm a Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) diagnosis of depression. The scale spans 0-5 to score "How much of the time..." with 0=at no time and 5=all the time; the higher the score, the more severe the depressive symptom.
Major Depression Inventory (MDI) | Day 30 of treatment intervention
  A brief (10-Item) behavioral survey for assessing clinical depression symptoms and severity; can confirm a DSM-IV diagnosis of depression. The scale spans 0-5 to score "How much of the time..." with 0=at no time and 5=all the time; the higher the score, the more severe the depressive symptom.
Major Depression Inventory (MDI) | Day 60 of treatment intervention
  A brief (10-Item) behavioral survey for assessing clinical depression symptoms and severity; can confirm a DSM-IV diagnosis of depression. The scale spans 0-5 to score "How much of the time..." with 0=at no time and 5=all the time; the higher the score, the more severe the depressive symptom.
Major Depression Inventory (MDI) | Day 1 of placebo intervention, before placebo consumption
  A brief (10-Item) behavioral survey for assessing clinical depression symptoms and severity; can confirm a DSM-IV diagnosis of depression. The scale spans 0-5 to score "How much of the time..." with 0=at no time and 5=all the time; the higher the score, the more severe the depressive symptom.
Major Depression Inventory (MDI) | Day 30 of placebo intervention
  A brief (10-Item) behavioral survey for assessing clinical depression symptoms and severity; can confirm a DSM-IV diagnosis of depression. The scale spans 0-5 to score "How much of the time..." with 0=at no time and 5=all the time; the higher the score, the more severe the depressive symptom.
Major Depression Inventory (MDI) | Day 60 of placebo intervention
  A brief (10-Item) behavioral survey for assessing clinical depression symptoms and severity; can confirm a DSM-IV diagnosis of depression. The scale spans 0-5 to score "How much of the time..." with 0=at no time, and 5=all the time; the higher the score, the more severe the depressive symptom.
Generalized Anxiety Disorder 7-item (GAD-7) scale | Day 1 of treatment intervention, before treatment consumption
  A brief behavioral scale for measuring symptoms related to general anxiety. The scale spans 0-3 to score the frequency of anxiety symptoms with 0=not at all sure and 3=nearly every day; the higher the score, the more frequent the anxiety symptom.
Generalized Anxiety Disorder 7-item (GAD-7) scale | Day 30 of treatment intervention
  A brief behavioral scale for measuring symptoms related to general anxiety. The scale spans 0-3 to score the frequency of anxiety symptoms with 0=not at all sure and 3=nearly every day; the higher the score, the more frequent the anxiety symptom.
Generalized Anxiety Disorder 7-item (GAD-7) scale | Day 60 of treatment intervention
  A brief behavioral scale for measuring symptoms related to general anxiety. The scale spans 0-3 to score the frequency of anxiety symptoms with 0=not at all sure and 3=nearly every day; the higher the score, the more frequent the anxiety symptom.
Generalized Anxiety Disorder 7-item (GAD-7) scale | Day 1 of placebo intervention, before placebo consumption
  A brief behavioral scale for measuring symptoms related to general anxiety. The scale spans 0-3 to score the frequency of anxiety symptoms with 0=not at all sure and 3=nearly every day; the higher the score, the more frequent the anxiety symptom.
Generalized Anxiety Disorder 7-item (GAD-7) scale | Day 30 of placebo intervention
  A brief behavioral scale for measuring symptoms related to general anxiety. The scale spans 0-3 to score the frequency of anxiety symptoms with 0=not at all sure and 3=nearly every day; the higher the score, the more frequent the anxiety symptom.
Generalized Anxiety Disorder 7-item (GAD-7) scale | Day 60 of placebo intervention
  A brief behavioral scale for measuring symptoms related to general anxiety. The scale spans 0-3 to score the frequency of anxiety symptoms with 0=not at all sure and 3=nearly every day; the higher the score, the more frequent the anxiety symptom.
Structured Interview Guide for the Hamilton Depression Scale and Inventory of Depressive Symptomatology-Clinician Rated (SIGHD-IDSC) | Day 1 of treatment intervention, before treatment consumption
  A verbal interview probing depressive symptoms based on two separate scales; the Hamilton Depression Scale and the Inventory of Depressive Symptomatology. Scores span 0-4 and are question-specific.
Structured Interview Guide for the Hamilton Depression Scale and Inventory of Depressive Symptomatology-Clinician Rated (SIGHD-IDSC) | Day 60 of treatment intervention
  A verbal interview probing depressive symptoms based on two separate scales; the Hamilton Depression Scale and the Inventory of Depressive Symptomatology. Scores span 0-4 and are question-specific.
Structured Interview Guide for the Hamilton Depression Scale and Inventory of Depressive Symptomatology-Clinician Rated (SIGHD-IDSC) | Day 1 of placebo intervention, before placebo consumption
  A verbal interview probing depressive symptoms based on two separate scales; the Hamilton Depression Scale and the Inventory of Depressive Symptomatology. Scores span 0-4 and are question-specific.
Structured Interview Guide for the Hamilton Depression Scale and Inventory of Depressive Symptomatology-Clinician Rated (SIGHD-IDSC) | Day 60 of placebo intervention
  A verbal interview probing depressive symptoms based on two separate scales; the Hamilton Depression Scale and the Inventory of Depressive Symptomatology. Scores span 0-4 and are question-specific.

SECONDARY OUTCOMES:
C-Reactive Protein (CRP) Measure | Immediately after enrollment, 30 days before start of intervention
  Biological measure of C-Reactive Protein from participant blood sample
CRP Measure | Day 1 of treatment intervention, before treatment consumption
  Biological measure of C-Reactive Protein from participant blood sample
CRP Measure | Day 30 of treatment intervention
  Biological measure of C-Reactive Protein from participant blood sample
CRP Measure | Day 60 of treatment intervention
  Biological measure of C-Reactive Protein from participant blood sample
CRP Measure | Day 1 of placebo intervention, before placebo consumption
  Biological measure of C-Reactive Protein from participant blood sample
CRP Measure | Day 30 of placebo intervention
  Biological measure of C-Reactive Protein from participant blood sample
CRP Measure | Day 60 of placebo intervention
  Biological measure of C-Reactive Protein from participant blood sample
Gut Microbiome Analysis | Day 1 of treatment intervention, before treatment consumption
  uBiome Explorer (TM) Microbiome Sampling Kit; tests microbial communities present in the gut microbiome
Gut Microbiome Analysis | Day 30 of treatment intervention
  uBiome Explorer (TM) Microbiome Sampling Kit; tests microbial communities present in the gut microbiome
Gut Microbiome Analysis | Day 60 of treatment intervention
  uBiome Explorer (TM) Microbiome Sampling Kit; tests microbial communities present in the gut microbiome
Gut Microbiome Analysis | Day 1 of placebo intervention, before placebo consumption
  uBiome Explorer (TM) Microbiome Sampling Kit; tests microbial communities present in the gut microbiome
Gut Microbiome Analysis | Day 30 of placebo intervention
  uBiome Explorer (TM) Microbiome Sampling Kit; tests microbial communities present in the gut microbiome
Gut Microbiome Analysis | Day 60 of placebo intervention
  uBiome Explorer (TM) Microbiome Sampling Kit; tests microbial communities present in the gut microbiome
Leeds Sleep Evaluation Questionnaire (LSEQ) | Day 1 of treatment intervention, before treatment consumption
  A short 10-item survey which probes issues related to sleep including falling asleep, quality and duration of sleep, and waking up after sleep. The scale for each of the 10 items is a line segment on which participants mark a tick; toward one end of the line is worse, toward the other end is better. A discrete datum is extracted from each continuous line by measuring to ticks from one end of the line with a ruler.
Leeds Sleep Evaluation Questionnaire (LSEQ) | Day 30 of treatment intervention
  A short 10-item survey which probes issues related to sleep including falling asleep, quality and duration of sleep, and waking up after sleep. The scale for each of the 10 items is a line segment on which participants mark a tick; toward one end of the line is worse, toward the other end is better. A discrete datum is extracted from each continuous line by measuring to ticks from one end of the line with a ruler.
Leeds Sleep Evaluation Questionnaire (LSEQ) | Day 60 of treatment intervention
  A short 10-item survey which probes issues related to sleep including falling asleep, quality and duration of sleep, and waking up after sleep. The scale for each of the 10 items is a line segment on which participants mark a tick; toward one end of the line is worse, toward the other end is better. A discrete datum is extracted from each continuous line by measuring to ticks from one end of the line with a ruler.
Leeds Sleep Evaluation Questionnaire (LSEQ) | Day 1 of placebo intervention, before placebo consumption
  A short 10-item survey which probes issues related to sleep including falling asleep, quality and duration of sleep, and waking up after sleep. The scale for each of the 10 items is a line segment on which participants mark a tick; toward one end of the line is worse, toward the other end is better. A discrete datum is extracted from each continuous line by measuring to ticks from one end of the line with a ruler.
Leeds Sleep Evaluation Questionnaire (LSEQ) | Day 30 of placebo intervention
  A short 10-item survey which probes issues related to sleep including falling asleep, quality and duration of sleep, and waking up after sleep. The scale for each of the 10 items is a line segment on which participants mark a tick; toward one end of the line is worse, toward the other end is better. A discrete datum is extracted from each continuous line by measuring to ticks from one end of the line with a ruler.
Leeds Sleep Evaluation Questionnaire (LSEQ) | Day 60 of placebo intervention
  A short 10-item survey which probes issues related to sleep including falling asleep, quality and duration of sleep, and waking up after sleep. The scale for each of the 10 items is a line segment on which participants mark a tick; toward one end of the line is worse, toward the other end is better. A discrete datum is extracted from each continuous line by measuring to ticks from one end of the line with a ruler.
Concentration of reactive oxygen species (ROS) | Day 1 of treatment intervention, before treatment consumption
  Electron paramagnetic resonance (EPR) to measures reactive oxygen species (ROS) in participant blood samples
Concentration of reactive oxygen species (ROS) | Day 30 of treatment intervention
  Electron paramagnetic resonance (EPR) measures reactive oxygen species (ROS) in participant blood samples
Concentration of reactive oxygen species (ROS) | Day 60 of treatment intervention
  Electron paramagnetic resonance (EPR) measures reactive oxygen species (ROS) in participant blood samples
Concentration of reactive oxygen species (ROS) | Day 1 of placebo intervention, before placebo consumption
  Electron paramagnetic resonance (EPR) measures reactive oxygen species (ROS) in participant blood samples
Concentration of reactive oxygen species (ROS) | Day 30 of placebo intervention
  Electron paramagnetic resonance (EPR) measures reactive oxygen species (ROS) in participant blood samples
Concentration of reactive oxygen species (ROS) | Day 60 of placebo intervention
  Electron paramagnetic resonance (EPR) measures reactive oxygen species (ROS) in participant blood samples
Concentration of quinolinic acid | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure quinolinic acid in participant blood samples
Concentration of quinolinic acid | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure quinolinic acid in participant blood samples
Concentration of quinolinic acid | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure quinolinic acid in participant blood samples
Concentration of quinolinic acid | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure quinolinic acid in participant blood samples
Concentration of quinolinic acid | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure quinolinic acid in participant blood samples
Concentration of quinolinic acid | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure quinolinic acid in participant blood samples
Concentration of kynurenic acid | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenic acid in participant blood samples
Concentration of kynurenic acid | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenic acid in participant blood samples
Concentration of kynurenic acid | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenic acid in participant blood samples
Concentration of kynurenic acid | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenic acid in participant blood samples
Concentration of kynurenic acid | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenic acid in participant blood samples
Concentration of kynurenic acid | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenic acid in participant blood samples
Concentration of kynurenine | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenine in participant blood samples
Concentration of kynurenine | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenine in participant blood samples
Concentration of kynurenine | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenine in participant blood samples
Concentration of kynurenine | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenine in participant blood samples
Concentration of kynurenine | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenine in participant blood samples
Concentration of kynurenine | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure kynurenine in participant blood samples
Concentration of tryptophan | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure tryptophan in participant blood samples
Concentration of tryptophan | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure tryptophan in participant blood samples
Concentration of tryptophan | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure tryptophan in participant blood samples
Concentration of tryptophan | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure tryptophan in participant blood samples
Concentration of tryptophan | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure tryptophan in participant blood samples
Concentration of tryptophan | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure tryptophan in participant blood samples
Concentration of indoleamine 2,3-dioxygenase (IDO) | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure indoleamine 2,3-dioxygenase (IDO) in participant blood samples
Concentration of indoleamine 2,3-dioxygenase (IDO) | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure indoleamine 2,3-dioxygenase (IDO) in participant blood samples
Concentration of indoleamine 2,3-dioxygenase (IDO) | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure indoleamine 2,3-dioxygenase (IDO) in participant blood samples
Concentration of indoleamine 2,3-dioxygenase (IDO) | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure indoleamine 2,3-dioxygenase (IDO) in participant blood samples
Concentration of indoleamine 2,3-dioxygenase (IDO) | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure indoleamine 2,3-dioxygenase (IDO) in participant blood samples
Concentration of indoleamine 2,3-dioxygenase (IDO) | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure indoleamine 2,3-dioxygenase (IDO) in participant blood samples
Concentration suicide-associated protein spindle and kinetochore-associated protein 2 (SKA-2) | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure SKA-2 in participant blood samples
Concentration of suicide-associated protein SKA-2 | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SKA-2 in participant blood samples
Concentration of suicide-associated protein SKA-2 | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SKA-2 in participant blood samples
Concentration of suicide-associated protein SKA-2 | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure SKA-2 in participant blood samples
Concentration of suicide-associated protein SKA-2 | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SKA-2 in participant blood samples
Concentration of suicide-associated protein SKA-2 | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SKA-2 in participant blood samples
Concentration of suicide-associated protein spermidine/spermine N1-acetyltransferase 1 (SAT-1) | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure SAT-1 in participant blood samples
Concentration of suicide-associated protein SAT-1 | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SAT-1 in participant blood samples
Concentration of suicide-associated protein SAT-1 | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SAT-1 in participant blood samples
Concentration of suicide-associated protein SAT-1 | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure SAT-1 in participant blood samples
Concentration of suicide-associated protein SAT-1 | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SAT-1 in participant blood samples
Concentration of suicide-associated protein SAT-1 | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SAT-1 in participant blood samples
Concentration of suicide-associated protein solute carrier family 4 member 4 (SLC4A4) | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure SLC4A4 in participant blood samples
Concentration of suicide-associated protein SLC4A4 | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SLC4A4 in participant blood samples
Concentration of suicide-associated protein SLC4A4 | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SLC4A4 in participant blood samples
Concentration of suicide-associated protein SLC4A4 | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure SLC4A4 in participant blood samples
Concentration of suicide-associated protein SLC4A4 | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SLC4A4 in participant blood samples
Concentration of suicide-associated protein SLC4A4 | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure SLC4A4 in participant blood samples
Concentration of brain-derived neurotropic factor (BDNF) | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure brain-derived neurotropic factor (BDNF) in participant plasma samples
Concentration of brain-derived neurotropic factor (BDNF) | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure brain-derived neurotropic factor (BDNF) in participant plasma samples
Concentration of brain-derived neurotropic factor (BDNF) | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure brain-derived neurotropic factor (BDNF) in participant plasma samples
Concentration of brain-derived neurotropic factor (BDNF) | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure brain-derived neurotropic factor (BDNF) in participant plasma samples
Concentration of brain-derived neurotropic factor (BDNF) | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure brain-derived neurotropic factor (BDNF) in participant plasma samples
Concentration of brain-derived neurotropic factor (BDNF) | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure brain-derived neurotropic factor (BDNF) in participant plasma samples
Concentration of glial cell line-derived neurotropic factor (GDNF) | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure glial cell line-derived neurotropic factor (GDNF) in participant plasma samples
Concentration of glial cell line-derived neurotropic factor (GDNF) | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure glial cell line-derived neurotropic factor (GDNF) in participant plasma samples
Concentration of glial cell line-derived neurotropic factor (GDNF) | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure glial cell line-derived neurotropic factor (GDNF) in participant plasma samples
Concentration of glial cell line-derived neurotropic factor (GDNF) | Day 1 of placebo intervention, before placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure glial cell line-derived neurotropic factor (GDNF) in participant plasma samples
Concentration of glial cell line-derived neurotropic factor (GDNF) | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure glial cell line-derived neurotropic factor (GDNF) in participant plasma samples
Concentration of glial cell line-derived neurotropic factor (GDNF) | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure glial cell line-derived neurotropic factor (GDNF) in participant plasma samples
Concentration of serotonin related compound serotonin transporter (SERT) | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure serotonin transporter (SERT) in participant blood samples
Concentration of serotonin related compound SERT | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure serotonin transporter (SERT) in participant blood samples
Concentration of serotonin related compound SERT | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure serotonin transporter (SERT) in participant blood samples
Concentration of serotonin related compound SERT | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure serotonin transporter (SERT) in participant blood samples
Concentration of serotonin related compound SERT | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure serotonin transporter (SERT) in participant blood samples
Concentration of serotonin related compound SERT | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure serotonin transporter (SERT) in participant blood samples
Concentration of serotonin related compound 5-hydroxyindoleacetic acid (5-HIAA) | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure 5-hydroxyindoleacetic acid (5-HIAA) in participant blood samples
Concentration of serotonin related compound 5-HIAA | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure 5-hydroxyindoleacetic acid (5-HIAA) in participant blood samples
Concentration of serotonin related compound 5-HIAA | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure 5-hydroxyindoleacetic acid (5-HIAA) in participant blood samples
Concentration of serotonin related compound 5-HIAA | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure 5-hydroxyindoleacetic acid (5-HIAA) in participant blood samples
Concentration of serotonin related compound 5-HIAA | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure 5-hydroxyindoleacetic acid (5-HIAA) in participant blood samples
Concentration of serotonin related compound 5-HIAA | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure 5-hydroxyindoleacetic acid (5-HIAA) in participant blood samples
Concentration of glutamate | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamate in participant blood samples
Concentration of glutamate | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamate in participant blood samples
Concentration of glutamate | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamate in participant blood samples
Concentration of glutamate | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamate in participant blood samples
Concentration of glutamate | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamate in participant blood samples
Concentration of glutamate | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamate in participant blood samples
Concentration of glutamine | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamine in participant blood samples
Concentration of glutamine | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamine in participant blood samples
Concentration of glutamine | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamine in participant blood samples
Concentration of glutamine | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamine in participant blood samples
Concentration of glutamine | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamine in participant blood samples
Concentration of glutamine | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of glutamine in participant blood samples
Concentration of cortisol | Day 1 of treatment intervention, before treatment consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of cortisol in participant blood samples
Concentration of cortisol | Day 30 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of cortisol in participant blood samples
Concentration of cortisol | Day 60 of treatment intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of cortisol in participant blood samples
Concentration of cortisol | Day 1 of placebo intervention, before placebo consumption
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of cortisol in participant blood samples
Concentration of cortisol | Day 30 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of cortisol in participant blood samples
Concentration of cortisol | Day 60 of placebo intervention
  Enzyme-linked immunosorbent assay (ELISA) to measure concentration of cortisol in participant blood samples
Concentration of inflammation biomarker interleukin 6 (IL-6) | Day 1 of treatment intervention, before treatment consumption
  Luminex assay to measure interleukin 6 (IL-6) in participant blood samples
Concentration of inflammation biomarker interleukin 6 (IL-6) | Day 30 of treatment intervention
  Luminex assay to measure interleukin 6 (IL-6) in participant blood samples
Concentration of inflammation biomarker interleukin 6 (IL-6) | Day 60 of treatment intervention
  Luminex assay to measure interleukin 6 (IL-6) in participant blood samples
Concentration of inflammation biomarker interleukin 6 (IL-6) | Day 1 of placebo intervention, before placebo consumption
  Luminex assay to measure interleukin 6 (IL-6) in participant blood samples
Concentration of inflammation biomarker interleukin 6 (IL-6) | Day 30 of placebo intervention
  Luminex assay to measure interleukin 6 (IL-6) in participant blood samples
Concentration of inflammation biomarker interleukin 6 (IL-6) | Day 60 of placebo intervention
  Luminex assay to measure interleukin 6 (IL-6) in participant blood samples
Concentration of inflammation biomarker interleukin 1 beta (IL-1beta) | Day 1 of treatment intervention, before treatment consumption
  Luminex assay to measure interleukin 1 beta (IL-1beta) in participant blood samples
Concentration of inflammation biomarker interleukin 1 beta (IL-1beta) | Day 30 of treatment intervention
  Luminex assay to measure interleukin 1 beta (IL-1beta) in participant blood samples
Concentration of inflammation biomarker interleukin 1 beta (IL-1beta) | Day 60 of treatment intervention
  Luminex assay to measure interleukin 1 beta (IL-1beta) in participant blood samples
Concentration of inflammation biomarker interleukin 1 beta (IL-1beta) | Day 1 of placebo intervention, before placebo consumption
  Luminex assay to measure interleukin 1 beta (IL-1beta) in participant blood samples
Concentration of inflammation biomarker interleukin 1 beta (IL-1beta) | Day 30 of placebo intervention
  Luminex assay to measure interleukin 1 beta (IL-1beta) in participant blood samples
Concentration of inflammation biomarker interleukin 1 beta (IL-1beta) | Day 60 of placebo intervention
  Luminex assay to measure interleukin 1 beta (IL-1beta) in participant blood samples
Concentration of inflammation biomarker interferon gamma (IFN-gamma) | Day 1 of treatment intervention, before treatment consumption
  Luminex assay to measure interferon gamma (IFN-gamma) in participant blood samples
Concentration of inflammation biomarker interferon gamma (IFN-gamma) | Day 30 of treatment intervention
  Luminex assay to measure interferon gamma (IFN-gamma) in participant blood samples
Concentration of inflammation biomarker interferon gamma (IFN-gamma) | Day 60 of treatment intervention
  Luminex assay to measure interferon gamma (IFN-gamma) in participant blood samples
Concentration of inflammation biomarker interferon gamma (IFN-gamma) | Day 1 of placebo intervention, before placebo consumption
  Luminex assay to measure interferon gamma (IFN-gamma) in participant blood samples
Concentration of inflammation biomarker interferon gamma (IFN-gamma) | Day 30 of placebo intervention
  Luminex assay to measure interferon gamma (IFN-gamma) in participant blood samples
Concentration of inflammation biomarker interferon gamma (IFN-gamma) | Day 60 of placebo intervention
  Luminex assay to measure interferon gamma (IFN-gamma) in participant blood samples
Concentration of inflammation biomarker tumour necrosis factor alpha (TNF-alpha) | Day 1 of treatment intervention, before treatment consumption
  Luminex assay to measure tumour necrosis factor alpha (TNF-alpha) in participant blood samples
Concentration of inflammation biomarker tumour necrosis factor alpha (TNF-alpha) | Day 30 of treatment intervention
  Luminex assay to measure tumour necrosis factor alpha (TNF-alpha) in participant blood samples
Concentration of inflammation biomarker tumour necrosis factor alpha (TNF-alpha) | Day 60 of treatment intervention
  Luminex assay to measure tumour necrosis factor alpha (TNF-alpha) in participant blood samples
Concentration of inflammation biomarker tumour necrosis factor alpha (TNF-alpha) | Day 1 of placebo intervention, before placebo consumption
  Luminex assay to measure tumour necrosis factor alpha (TNF-alpha) in participant blood samples
Concentration of inflammation biomarker tumour necrosis factor alpha (TNF-alpha) | Day 30 of placebo intervention
  Luminex assay to measure tumour necrosis factor alpha (TNF-alpha) in participant blood samples
Concentration of inflammation biomarker tumour necrosis factor alpha (TNF-alpha) | Day 60 of placebo intervention
  Luminex assay to measure tumour necrosis factor alpha (TNF-alpha) in participant blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Francis, Ph.D., Principal Investigator — Louisiana State University, Baton Rouge
Locations (2):
- United States (2):
  - Cottonport Family Clinic, Cottonport, Louisiana
  - Marksville Family Clinic, Marksville, Louisiana

IPD SHARING:
Plan to Share IPD: No